CLINICAL TRIAL: NCT05230056
Title: Effectiveness and Therapeutic Compliance of Digital Therapy in Shoulder Rehabilitation.
Brief Title: Digital Therapy in Shoulder Rehabilitation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLYDT
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PG (Experimental)
  Interventions: Behavioral: PG
- CTRL (Active Comparator)
  Interventions: Behavioral: CTRL

INTERVENTIONS:
Behavioral: PG — Shoulder Digital therapy
  Arms: PG
Behavioral: CTRL — Shoulder non-digital therapy
  Arms: CTRL

SUMMARY:
Digital therapy may provides real time visual feedbacks. Instrumented devices objectively quantify the patient's performance during rehabilitation and thus could be helpful for the personalization of the exercises.

The interactive ball of this trial allows measuring both movement and pressure applied on it. Therefore, the objectives of this study are: (i) to evaluate whether the use of a novel digital therapy gaming system was therapeutically relevant during shoulder rehabilitation; (ii) to understand whether the device was effective in improving patients' engagement in comparison to a control non-gaming rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* impingement syndrome, capsulitis, tendon injuries, degenerative joint or tendon pathologies
* pain between 2/10 and 8/10 on a visual analogue scale

Exclusion Criteria:

* post-surgical patients
* inability to perform active exercises
* peripheral neurological deficits
* cervical-brachialgia
* algodystrophy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
shoulder pain | From baseline up to two weeks
  Shoulder pain by means of Visual Analogue Scale (no pain:0; maximal pain: 10)
shoulder strength | From baseline up to two weeks
  Shoulder strength by means of an isometric maximal voluntary contraction measured in kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rizzato A, Pizzichemi M, Gobbi E, Gerardi A, Fortin C, Copcia A, Paoli A, Marcolin G. Effectiveness and therapeutic compliance of digital therapy in shoulder rehabilitation: a randomized controlled trial. J Neuroeng Rehabil. 2023 Jul 8;20(1):87. doi: 10.1186/s12984-023-01188-7. PMID 37420268